CLINICAL TRIAL: NCT02946931
Title: The Drug Use-results Survey (All-Case Surveillance) on Prizbind® for Intravenous Solution 2.5 g in Japan
Brief Title: All-Case Surveillance of Prizbind®
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1321.15
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — idarucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Prizbind® for Intravenous Solution: Patients treated with dabigatran etexilate who have uncontrolled bleeding or require emergency surgery or procedures.
  Interventions: Drug: Prizbind®

INTERVENTIONS:
Drug: Prizbind® — Prizbind®
  Other Names: Idarucizumab

SUMMARY:
To evaluate safety and effectiveness of Prizbind® for Intravenous Solution 2.5 g under Japanese clinical condition.

ELIGIBILITY:
Inclusion criteria:

Patients who are prescribed with Prizbind® for Intravenous Solution 2.5 g by the discretion of investigators

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are prescribed with Prizbind
Sampling Method: Non-Probability Sample
Enrollment: 1402 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Yasaka M, Yokota H, Suzuki M, Asakura H, Yamane T, Ogi Y, Kimoto T, Nakayama D. Idarucizumab for Emergency Reversal of the Anticoagulant Effects of Dabigatran: Final Results of a Japanese Postmarketing Surveillance Study. Cardiol Ther. 2023 Dec;12(4):723-740. doi: 10.1007/s40119-023-00333-6. Epub 2023 Oct 17. PMID 37845427
- [Derived] Yasaka M, Yokota H, Suzuki M, Asakura H, Yamane T, Ogi Y, Ochiai K, Nakayama D. Idarucizumab for Emergency Reversal of Anticoagulant Effects of Dabigatran: Interim Results of a Japanese Post-Marketing Surveillance Study. Cardiol Ther. 2020 Jun;9(1):167-188. doi: 10.1007/s40119-020-00165-8. Epub 2020 Mar 9. PMID 32152956
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This post marketing surveillance (PMS) was a non-interventional study based on new data collection to gather data on safety and effectiveness of the Prizbind® for Intravenous Solution under Japanese clinical condition. All patients were administered Prizbind® for Intravenous Solution after the approval at the sites contracted with the sponsor were to be registered.
Pre-assignment Details: All patients who are prescribed with Prizbind® for Intravenous Solution 2.5 g by the discretion of investigators were enrolled. Any screening was not conducted.
Groups:
- Prizbind® for Intravenous Solution: Patients who had been treated with dabigatran etexilate and required rapid reversal of the anticoagulant effects of dabigatran were administered intravenously 2 vials of 2.5 gram (g) of Prizbind® (total dose: 5 g). Two vials of Prizbind® were administered as two consecutive infusions over 5 to 10 minutes each or as a bolus injection.
Period: Overall Study
Arm/Group | Prizbind® for Intravenous Solution
Started (Treated with Prizbind®) | 1402
Case Report Forms (CRFs) Collected | 814
CRFs Valid | 813
Completed | 571
Not Completed | 831
Not completed — Did not require collection of CRFs | 588
Not completed — Other than listed | 37
Not completed — Discharge from hospital | 118
Not completed — Adverse Event | 81
Not completed — CRFs not valid | 1
Not completed — CRFs with missing information on the date of termination of PMS | 6

BASELINE CHARACTERISTICS:
Population: Safety Set: This patient set included all patients who had no invalid registration, who were documented to have taken at least one dose of Prizbind®.
Arm/Group | Prizbind® for Intravenous Solution
Number analyzed (Participants) | 813
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267
  Male | 546
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Drug Reactions (ADRs)
Description: Adverse reaction was defined as a response to the medicinal product which was noxious and unintended. Number of participants with Adverse Drug Reactions (ADRs) is reported.
Time Frame: From the first intake of Prizbind® for Intravenous Solution 2.5 g to the end of the observation period for each patient, up to 74 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Prizbind® for Intravenous Solution
Number analyzed (Participants) | 813
Participants | 30

2. Secondary Outcome: Maximum Reversal of Anticoagulation as Measured by Activated Partial Thromboplastin Time (aPTT)
Description: Maximum reversal of anticoagulation as measured by activated partial thromboplastin time (aPTT) is reported.
  Maximum reversal was calculated as:｛(predose aPTT - minimum postdose aPTT)/(predose aPTT - upper limit of normal (ULN))｝ × 100%. If calculated reversal is > 100, it was set to 100.
Time Frame: From the end of the first infusion up to 4 hours after the last infusion on Day 1.
Population: Patients of the effectiveness set (all patients with Prizbind® in the safety set who have at least one available effectiveness data) whose activated partial thromboplastin time (aPTT) value at baseline exceeded the upper limit of normal (ULN).
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Prizbind® for Intravenous Solution
Number analyzed (Participants) | 103
percentage | 100.0 [82.50 to 100.0]

3. Secondary Outcome: Number of Patients in Each Category of Maximum Reversal of Anticoagulation as Measured by Activated Partial Thromboplastin Time (aPTT)
Description: Number of patients in each category of maximum reversal of anticoagulation as measured by activated partial thromboplastin time (aPTT) is reported.
  Maximum reversal was calculated as:｛(predose aPTT - minimum postdose aPTT)/(predose aPTT - upper limit of normal (ULN))｝ × 100%. If calculated reversal is > 100, it was set to 100.
  Maximum Reversal was categorized in the following 4 categories:
  100% 80% <= and < 100% 50% <= and < 80% < 50%
Time Frame: From the end of the first infusion up to 4 hours after the last infusion on Day 1.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Prizbind® for Intravenous Solution
Number analyzed (Participants) | 103
Participants
  100 % | 65
  80<= and <100 % | 16
  50<= and <80 % | 9
  <50 % | 13

ADVERSE EVENTS:
Time Frame: From the first intake of Prizbind® for Intravenous Solution 2.5 g to the end of the observation period for each patient, up to 74 days.
Description: Safety Set: This patient set included all patients who had no invalid registration, who were documented to have taken at least one dose of Prizbind®.
Arm/Group | Prizbind® for Intravenous Solution
All-Cause Mortality (participants affected / at risk) | 103/813
Serious Adverse Events (participants affected / at risk) | 192/813
Other Adverse Events (participants affected / at risk) | 0/813
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prizbind® for Intravenous Solution (N=813)
Peritonitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Gangrene (Infections and infestations) | 1
Mediastinitis (Infections and infestations) | 1
Meningitis bacterial (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Systemic candida (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Delirium (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 16
Cerebral haemorrhage (Nervous system disorders) | 10
Brain oedema (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 5
Embolic stroke (Nervous system disorders) | 4
Epilepsy (Nervous system disorders) | 5
Cerebellar haemorrhage (Nervous system disorders) | 3
Haemorrhage intracranial (Nervous system disorders) | 2
Hydrocephalus (Nervous system disorders) | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2
Brain stem haemorrhage (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Spinal cord haemorrhage (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Vascular parkinsonism (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Eye haematoma (Eye disorders) | 1
Cardiac failure (Cardiac disorders) | 6
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericardial haemorrhage (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricle rupture (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Cardiac perforation (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Shock haemorrhagic (Vascular disorders) | 7
Haemorrhage (Vascular disorders) | 5
Arterial occlusive disease (Vascular disorders) | 3
Aortic dissection (Vascular disorders) | 2
Circulatory collapse (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Shock (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Arteriovenous fistula (Vascular disorders) | 1
Haemorrhagic infarction (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
Peripheral circulatory failure (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Coeliac artery occlusion (Vascular disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 5
Death (General disorders) | 3
Oedema (General disorders) | 1
Blood pressure decreased (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 19
Brain herniation (Injury, poisoning and procedural complications) | 4
Extradural haematoma (Injury, poisoning and procedural complications) | 4
Road traffic accident (Injury, poisoning and procedural complications) | 2
Brain contusion (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1
Postoperative delirium (Injury, poisoning and procedural complications) | 1
Pneumonia aspiration (Infections and infestations) | 20
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Aneurysm ruptured (Vascular disorders) | 1
Microscopic polyangiitis (Vascular disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 2
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Traumatic shock (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT02946931/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02946931/SAP_001.pdf